CLINICAL TRIAL: NCT01061398
Title: CT-FIRST: Cardiac Computed Tomography Versus Stress Imaging For Initial Risk STratification
Acronym: CT-FIRST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Todd C. Villines, Director, Cardiovascular Research, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WU#08-12032
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease; Chest Pain; Coronary Atherosclerosis; Stress Testing
Keywords: cardiac ct; stress testing; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac CT Arm (Experimental): Patients referred for stress imaging due to complaints consistent with possible angina, randomized to receive an additional cardiac CT scan.
  Interventions: Procedure: Cardiac CT Angiography
- No CT Arm (Active Comparator): Patients with symptoms consistent with possible angina, randomized to receive the type of stress imaging test ordered by their physician.
  Interventions: Procedure: Stress Imaging Test (Stress Myocardial Perfusion Study or Stress Echocardiogram)

INTERVENTIONS:
Procedure: Cardiac CT Angiography — Patients randomized to CT Arm will undergo 64-slice cardiac CT angiography (single scan) in addition to the stress imaging test ordered by their physician
  Arms: Cardiac CT Arm
Procedure: Stress Imaging Test (Stress Myocardial Perfusion Study or Stress Echocardiogram) — Stress imaging test as ordered by the subjects provider without option for cardiac CT angiography (no CT arm)
  Arms: No CT Arm

SUMMARY:
In patients with chest pain or shortness of breath who are referred for stress imaging tests (either stress echocardiography or stress nuclear testing), the investigators seek to compare impact of using cardiac CT scans of the heart arteries to the stress test that their doctors ordered.

DETAILED DESCRIPTION:
The current evaluation for chest pain in low and intermediate risk patients typically starts with a functional assessment for coronary ischemia. Exercise treadmill testing is often selected as the initial diagnostic modality for coronary artery function. However, exercise treadmill testing is limited by its modest sensitivity and specificity, often resulting in further cardiac resource utilization for patient risk stratification and reassurance. Additionally, many patients with chest pain are not candidates for regular stress testing due to an abnormal baseline electrocardiogram or inability to exercise. Therefore, exercise or pharmacologic stress imaging is considered the standard of care for the evaluation of coronary artery function in a large percentage of patients with chest pain. However, each of the currently available stress imaging tests has well-documented limitations, resulting in a sizeable number of false negative and false positive studies. With the advent of coronary Multislice Computed Tomography (MSCT) angiography, coronary artery anatomy can now be accurately evaluated noninvasively. Despite its impressive performance characteristics, the role of coronary MSCT angiography in the evaluation of angina remains undefined. Furthermore, studies comparing MSCT to stress imaging are lacking. CT-FIRST compares the impact on downstream resource utilization and patient outcomes of an initial diagnostic strategy employing the addition of coronary MSCT angiography to stress imaging (exercise and pharmacologic stress echo and nuclear perfusion testing) with a standard-of-care diagnostic strategy of stress imaging for the evaluation of low-intermediate risk patients with possible angina. The study is a single center, prospective, non-blinded, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years of age at time of enrollment.
* Chest pain or anginal equivalent symptoms possibly suggestive of symptomatic coronary artery disease
* Low-intermediate risk (<75% pretest probability) for symptomatic coronary artery disease on basis of age, sex, and quality of reported symptom as classified by the Diamond and Forrester scheme.
* Referred for a either a stress echocardiogram or a nuclear stress perfusion study.
* Ability to provide informed consent.

Exclusion Criteria:

* Presence of known pre-existing coronary artery disease (known prior myocardial infarction, ECG evidence of prior infarction, prior angiographic evidence of significant coronary artery disease, history of prior coronary revascularization).
* Previous outpatient or inpatient evaluation for coronary artery disease to include exercise treadmill testing, stress echocardiography or nuclear myocardial perfusion studies within the last 24 months.
* Presence of signs or symptoms that are clearly compatible with non-cardiac chest pain, including musculoskeletal, gastrointestinal or neuropathic causes.
* Renal insufficiency (creatinine >1.5mg/dl) or renal failure requiring dialysis.
* Baseline heart rate > 100bpm, atrial fibrillation or other markedly irregular rhythm (frequent ectopy, multifocal atrial tachycardia) on baseline ECG.
* Pregnancy or unknown pregnancy status.
* Known allergy to iodinated contrast.
* Inability to tolerate beta-blocking drugs, including patients with reactive airways disease requiring maintenance inhaled bronchodilators or steroids, complete heart block or second-degree atrioventricular block.
* Patients with hyperthyroidism including Grave's disease and toxic multinodular goiter
* Computed tomography imaging or iodinated contrast administration over 50 ml, within the past 48 hours.
* Inability to withhold ingestion of metformin or commonly used erectile dysfunction medications (Viagra, Cialis, Levitra) for 48 hours prior to and following MSCT scan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Rates of adverse cardiac events and resource utilization (rates of additional diagnostic tests that are performed for the initial complaint of angina/angina equivalent and clinical outpatient/inpatient/ED encounters for the initial cardiac complaint) | 24 months

SECONDARY OUTCOMES:
Total number and per-patient rates of adverse cardiac events (cardiac death, myocardial infarction, unstable angina, coronary revascularization) | 24 months
Total number and per-patient rates of subsequent cardiac diagnostic tests performed (stress tests, cardiac catheterizations, other tests) for the initial complaint of angina/angina equivalent | 24 months
Total number and per-patient rates of subsequent outpatient + inpatient + emergency department encounters for the initial cardiac complaint | 24 months
Avoidance of unnecessary cardiac catheterizations. An unnecessary cardiac catheterization is defined as a catheterization showing non-obstructive coronary disease and no cause for the symptoms. | 24 months
Change in motivation for healthy behavioral change | 24 months
Change in subject anxiety, as assessed by the State and Trait Anxiety Inventory | 24 months
Change in subject depression | 24 months
Satisfaction with diagnostic evaluation for initial complaint. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd C. Villines, M.D., Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States